CLINICAL TRIAL: NCT00934193
Title: Does Peri-Operative Gabapentin Reduce Chronic Post-Thoracotomy Pain?
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Wichita Medical Research and Education Foundation (Other); Ascension Via Christi Hospitals Wichita, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 220081131; WMREF 80104-257 (Other: WMREF IRB)
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Post-thoracotomy Pain
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Gabapentin (Active Comparator)
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Treatment will consist of a 600 mg dose of gabapentin or placebo given preoperatively the night before surgery, based on a computer generated randomized assignment. The treatment group will continue to be medicated with gabapentin 300 mg twice daily for one month following surgery. Those not included in the treatment arm of the study will continue to take a placebo for the same duration. Follow-up will consist of a postoperative visit at approximately 48 hours and a one month clinical visit.
  Arms: Gabapentin
Drug: Placebo — Treatment will consist of a 600 mg dose of gabapentin or placebo given preoperatively the night before surgery, based on a computer generated randomized assignment. The treatment group will continue to be medicated with gabapentin 300 mg twice daily for one month following surgery. Those not included in the treatment arm of the study will continue to take a placebo for the same duration. Follow-up will consist of a postoperative visit at approximately 48 hours and a one month clinical visit.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine if gabapentin can decrease or prevent chronic post-thoracotomy pain.

DETAILED DESCRIPTION:
This study is a prospective double blind randomized controlled trial evaluating the peri-operative use of gabapentin in the prevention or modulation of post-thoracotomy hyperalgesia. Treatment will consist of a 600 mg dose of gabapentin or placebo given preoperatively the night before surgery, based on a computer generated randomized assignment. The treatment group will continue to be medicated with gabapentin 300 mg twice daily for one month following surgery. Those not included in the treatment arm of the study will continue to take a placebo for the same duration. Follow-up will consist of a postoperative visit at approximately 48 hours and a one month clinical visit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Undergoing non-cardiac thoracic surgeries
* Patients determined to have impaired decisional capacity with respect to the provision of informed consent or prisoners will not be included in the study.

Exclusion Criteria:

* Current gabapentin use or current treatment for neuropathic pain.
* Pregnant or considering becoming pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine if gabapentin can decrease or prevent chronic post-thoracotomy pain. | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Sinisa Malinovic, MD, Principal Investigator — Ascension Via Christi Hospitals Wichita, Inc.